CLINICAL TRIAL: NCT02062203
Title: A Phase 1, Single-Center, Partially Double-Blinded, Active and Placebo Controlled, Randomized 4-Way Crossover Study to Evaluate the Effect of AKB-6548 on Cardiac Repolarization Intervals in Healthy Volunteers
Brief Title: Effect of AKB-6548 on Cardiac Repolarization Intervals in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AKB-6548-CI-0010
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Akebia; QT interval; TQT; pharmacokinetic; anemia; chronic kidney disease; CKD; chronic renal insufficiency; renal impairment; safety
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AKB-6548 (therapeutic dose) (Experimental)
  Interventions: Drug: AKB-6548 (therapeutic dose)
- AKB-6548 (supratherapeutic dose) (Experimental)
  Interventions: Drug: AKB-6548 (supratherapeutic dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: AKB-6548 (therapeutic dose) — Single oral dose of AKB-6548 at a therapeutic dose level
  Arms: AKB-6548 (therapeutic dose)
Drug: AKB-6548 (supratherapeutic dose) — Single oral dose of AKB-6548 at a supratherapeutic dose level
  Arms: AKB-6548 (supratherapeutic dose)
Drug: Placebo — Single oral dose of placebo
  Arms: Placebo
Drug: Moxifloxacin — Single oral dose of 400 mg moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
The main purpose of this study is to evaluate the effect of single oral therapeutic and supratherapeutic doses of AKB-6548 on the QT interval.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, non-smoking males or females, 18 and 55 years of age, inclusive
* BMI 18.0 and 32.0 kg/m2, inclusive
* non clinically significant 12-lead ECG
* heart rate of 45 to 90 beats per minute, inclusive
* mean systolic blood pressure <141 mmHg and mean diastolic blood pressure < 90 mmHg

Key Exclusion Criteria:

* history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, GI, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias, or torsades de pointes, structural heart disease, or a family history of Long QT syndrome
* significant abnormalities in liver function tests
* history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* history of Gilbert's Syndrome
* positive hepatitis panel
* seizure disorder or receiving anti-epilepsy medication for seizure disorder
* any acute or chronic condition that, in the opinion of the Investigator, may pose a safety risk to a subject in this study or which would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change-from-baseline QTcF (ΔΔQTcF) following AKB-6548 administration. | multiple timepoint evaluations from pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
Placebo-corrected change-from-baseline heart rate (HR), PR interval, QRS interval | multiple timepoint evaluations from pre-dose to 24 hours post-dose
Categorical outliers defined as QTcF >450 msec, 480 msec and 500 msec at any timepoint and change-from-baseline QTcF (ΔQTcF) >30 msec (increased by 30 msec) and >60 msec | multiple timepoint evaluations from pre-dose to 24 hours post-dose
Categorical outliers for HR, PR interval, QRS interval | multiple timepoint evaluations from pre-dose to 24 hours post-dose
Frequency of T wave morphology changes | multiple timepoint evaluations from pre-dose to 24 hours post-dose
Placebo-corrected change-from-baseline QTcF (ΔΔQTcF) following moxifloxacin administration | multiple timepoint evaluations from pre-dose to 24 hours post-dose
Safety parameters to include adverse events; changes in routine clinical laboratory measures including chemistry, hematology, and urinalysis; and clinically significant changes noted during physical examinations or in vital signs | from first dose of study medication through the final protocol required visit

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided